CLINICAL TRIAL: NCT05364671
Title: Multicenter Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Efficacy and Safety of Raphamin in the Treatment of Coronavirus Disease 2019 in Outpatients
Brief Title: Clinical Trial of Efficacy and Safety of Raphamin in the Treatment of Coronavirus Disease 2019 in Outpatients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-006
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2023-08

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raphamin (Experimental): Tablet for oral use.
  Interventions: Drug: Raphamin
- Placebo (Placebo Comparator): Tablet for oral use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raphamin — Tablet for oral use. The drug is administered not during meals. The tablet should be held in mouth until complete dissolution. On the first day, 8 tablets should be administered using the following regimen: 1 tablet every 30 minutes in the first 2 hours (5 tablets in total within 2 hours), then additionally one tablet 3 times with regular time intervals. From day 2 onwards, 1 tablet taken 3 times daily. The treatment period is 5 days.
  Other Names: MMH-407
  Arms: Raphamin
Drug: Placebo — Tablet for oral use. The drug is administered not during meals. The tablet should be held in mouth until complete dissolution. Placebo is administered according to the Raphamin regimen.
  Arms: Placebo

SUMMARY:
Multicenter double-blind placebo-controlled parallel-group randomized clinical trial of efficacy and safety of Raphamin in the treatment of coronavirus disease 2019 in outpatients.

DETAILED DESCRIPTION:
Design: multicenter, double blind, placebo-controlled, parallel group randomized clinical trial.

The study enrolls outpatients of either gender aged 18-75 years with increased body temperature > 37.5°C and other upper respiratory infection symptoms (cough, chest congestion, sore throat, nasal congestion/moderate rhinorrhea). The investigator should specify the patient's status of vaccination for COVID-19, influenza and other infections. Patients within the first four weeks after any vaccination/booster vaccination are not considered as candidates to participate in the study.

Nasopharyngeal swabs and rapid COVID-19 test are made after signing informed consent (two versions are used: 1) for patients consented for laboratory tests; 2) for patients without the consent).

Patients with a positive rapid test and presence of mild COVID-19 (upper respiratory infection symptoms, no symptoms of moderate or severe forms) within 24 hours after manifestation of the first disease symptoms are considered as candidates for the study. Oxygen saturation (SpO2) is measured by pulse oximetry in all patients (pulse oximeters are provided by the study sponsor). If SpO2 is ≥95%, a patient may be selected for the study. Baseline severity for COVID-19 symptoms is evaluated using the scoring system "Assessment of 14 Common COVID-19-Related Symptoms" (FDA, 2020). This scoring system assesses the follows symptoms:

1. Stuffy or runny nose.
2. Sore throat.
3. Shortness of breath (difficulty breathing).
4. Cough.
5. Low energy or tiredness.
6. Muscle or body aches.
7. Headache.
8. Chills or shivering.
9. Feeling hot or feverish.
10. Nausea (feeling like you wanted to throw up).
11. Vomiting.
12. Diarrhea.
13. Sense of smell.
14. Sense of taste.

Each symptom is scored individually using the following scoring values:

* Items 1-10: None = 0; Mild = 1; Moderate = 2; and Severe = 3;
* Items 11 and 12: Not at all = 0; 1-2 times = 1; 3-4 times = 2; 5 or more times = 3;
* Items 13 and 14: Sense of smell/taste same as usual = 0; Sense of smell/taste less than usual = 1; No sense of smell/taste = 2.

The minimal baseline score for COVID-19-related symptoms is defined as follows: at least two symptoms with a score of 2 or higher, with the exception of taste and smell where subjects may have a score of 1 or higher, and the absence of shortness of breath (difficulty breathing).

If more severe symptoms are presented, the patient is not included in the study. The therapeutic approach is determined by the current edition of the clinical recommendations of the Ministry of Health of the Russian Federation "Prevention, diagnosis and treatment of a new coronavirus infection (COVID-19)".

At visit 1 (Day 1), in addition to rapid COVID-19 test and SpO2 measurement, the investigator will collect complaints and medical history of the patient, perform objective examination including vital signs (blood pressure, heart rate and respiration rate), record concomitant diseases and concomitant therapy, perform nasopharyngeal smearing for further PCR for SARS-CoV-2, laboratory tests will be made (if the patient gave his/her consent for blood and urine sampling).

Patients who meet all the inclusion criteria and do not have exclusion criteria at Visit 1 (Day 1) are randomized into one of two groups: patients in group 1 receive Raphamin for 5 days; patients in group 2 receive placebo according to the Raphamin regimen.

If positive PCR test is received (confirmation of new coronavirus disease COVID-19), the patient continues to participate in the study. If PCR result is negative, the patient completes participation in the study ahead of schedule, and his further therapy is determined by the investigator in accordance with the standard of care.

Electronic patient diary (EPD) is utilized in the study where morning and evening axillary temperature records are made with the time of measurement. The sponsor provides a classical mercury-free thermometer to each patient. In addition, presence and severity of the disease symptoms according to the scoring system "Assessment of 14 Common COVID-19-Related Symptoms", antipyretics administration and probable worsening of disease duration should also be recorded in EPD. All patients are provided with paracetamol. The physician instructs the patient how to fill in the diary. The EPD is available for filling in within 28 days of participation in the study.

Overall, patients are observed for 28 days (screening and randomization up to 1 day, treatment for 5 days, follow-up till 28th day).

During the study, six visits are planned: on days 1, 3, 6, 10, 21, and 28 (visits 1, 2, 3, 4, 5, and 6). Visits 1, 3, and 4 are in person (visits to the patient or visits to the medical center) when the physician examines the patient and monitors EPD records. At visit 3, the patient's adherence to treatment is assessed and laboratory tests are performed. Visits 2, 5 and 6 are phone surveys to determine the patient's condition, presence/absence of complaints. In case of worsening of disease duration, the physician makes an extra visit. Patients with COVID-19 progression to more severe form as well as hospitalized patients are considered as reaching the study endpoints and terminate participation in the study ahead of schedule. The therapeutic approach is determined by the current edition of the clinical recommendations of the Ministry of Health of the Russian Federation "Prevention, diagnosis and treatment of a new coronavirus infection (COVID-19)".

During the study, the use of paracetamol and medicines for the treatment of concomitant diseases is allowed, with the exception of the drugs specified in the section "Prohibited concomitant treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-75 years old.
2. Diagnosis of new coronavirus infection COVID-19 based on medical examination: axillary temperature >37.5°C, upper respiratory infection symptoms, SpO2 ≥ 95%, no symptoms of moderate or severe forms.
3. The minimal baseline score for COVID-19-related symptoms defined as follows: at least two symptoms with a score of 2 or higher, with the exception of taste and smell where subjects may have a score of 1 or higher, and the absence of shortness of breath (difficulty breathing).
4. Positive rapid test for for SARS-CoV-2 (COVID-19).
5. The first 24 hours from the disease onset.
6. Patients giving their consent to use reliable contraception during the study.
7. Signed patient information sheet (informed consent form).

Exclusion Criteria:

1. Moderate and severe COVID-19.
2. The first four weeks after any vaccination/revaccination, including against COVID-19, influenza, pneumococcal and other infections.
3. Suspected pneumonia, bacterial infection (including otitis media, sinusitis, urinary tract infection, meningitis, sepsis, etc.).
4. Patients requiring medications prohibited within the study.
5. Medical history or previously diagnosed primary and secondary immunodeficiency.
6. Medical history/suspicion of oncology of any localization (except for benign neoplasms).
7. Exacerbation or decompensation of chronic diseases affecting the patient's ability to participate in the clinical study.
8. Malabsorption syndrome, including congenital or acquired lactase or disaccharidase deficiency, galactosemia.
9. Allergy/ hypersensitivity to any of the components of the medications used in the treatment.
10. Pregnancy, breast-feeding; childbirth less than 3 months prior to the inclusion in the trial, unwillingness to use contraceptive methods during the trial.
11. Use of medications listed in "Prohibited concomitant therapy" within 4 weeks before the study entry.
12. Patients who, from the investigator's point of view, will fail to comply with the requirements of the trial or with the intake regimen of the study drugs.
13. Medical history of mental diseases, alcoholism or drug abuse which, according to the investigator's opinion, will interfere with the study procedures.
14. Participation in other clinical trials within 3 months prior to enrollment in this study.
15. The patient is related to the study center staff directly involved in the trial or is the immediate relative of the investigator. Immediate family is defined as a spouse, parents, children or siblings, whether natural or adopted.
16. The patient works for OOO "NPF "MATERIA MEDICA HOLDING" i.e. is the company's employee, part-time employee under contract or appointed official in charge of the trial, or their immediate family.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- Russia (36):
  - Belgorod State National Research University, Department of Hospital Therapy, Belgorod
  - Ivanovo clinical hospital named after Kuvaevs/Polyclinic #10, Ivanovo
  - Kazan State Medical University, Department of Propedeutics of Internal Diseases named after prof. S.S. Zimnitsky, Kazan'
  - Kazan State Medical University/Department of Infectious Diseases, Kazan'
  - Kirov State Medical University, Hospital Therapy Department, Kirov
  - Kuban State Medical University, Infectious Diseases and Phthisiopulmonology, Krasnodar
  - Clinical hospital "RZD-Medicine" of the city of Nizhny Novgorod, Nizhny Novgorod
  - City Clinical Hospital # 2, Novosibirsk
  - Clinical Hospital # 4, Penza
  - LLC "Professor's Clinic", Perm
  - LLC "Ultrasound Clinic 4D", Pyatigorsk
  - Ryazan State Medical University named after Academician I.P. Pavlova, Ryazan
  - LLC "BioTechService", Saint Petersburg
  - City clinic # 44, Saint Petersburg
  - City Polyclinic # 25 of the Nevsky District, Saint Petersburg
  - LLC "Energy of Health", Saint Petersburg
  - LLC "Strategic medical systems", Saint Petersburg
  - Llc "Medical Clinic", Saint Petersburg
  - LLC "Research Center Eco-safety", Saint Petersburg
  - JSC "North-West Center for Evidence-Based Medicine", Saint Petersburg
  - LLC "Clinic Zvezdnaya", Saint Petersburg
  - City Polyclinic # 43, Saint Petersburg
  - Lomonosov Interdistrict Hospital named after I.N. Yudchenko, Saint Petersburg
  - City Intercession Hospital, Saint Petersburg
  - LLC "Meili", Saint Petersburg
  - City polyclinic # 74, Saint Petersburg
  - Samara City Hospital # 4, Samara
  - LLC "Center for DNA Research", Saratov
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - LLC "Scientific Medical Center for General Therapy and Pharmacology", Stavropol
  - Tver State Medical University, Tver'
  - Bashkir State Medical University, Internal Medicine Department, Ufa
  - Voronezh Regional Clinical Hospital # 1, Voronezh
  - Central city hospital, Yaroslavl
  - LLC "Medical Center for Diagnostics and Prevention Plus", Yaroslavl
  - Central city hospital # 7, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raphamin | Placebo
Started | 382 | 389
Completed | 356 | 358
Not Completed | 26 | 31
Not completed — Negative PCR result for SARS-CoV-2 | 20 | 26
Not completed — Patient's inability or refusal to comply with protocol requirements | 3 | 1
Not completed — Need to prescribe prohibited drugs in this study | 1 | 3
Not completed — Patient's desire to complete the study early due to treatment failure or any other reason | 2 | 0
Not completed — Deviation from the schedule of face-to-face visits on more than 1 day | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raphamin | Placebo | Total
Number analyzed (Participants) | 382 | 389 | 771
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 336 | 352 | 688
  >=65 years | 43 | 35 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (15.3) | 43.4 (14.3) | 43.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 249 | 482
  Male | 149 | 140 | 289
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 382 | 389 | 771

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With COVID-19 Progression to a More Severe Form
Description: Severity of COVID-19 is assessed in accordance with criteria presented in the current edition of the clinical recommendations of the Ministry of Health of the Russian Federation "Prevention, diagnosis and treatment of a new coronavirus infection (COVID-19)".
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
Participants | 59 | 89
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.0088, Chi-squared — A priori threshold for statistical significance is set to 0.04

2. Secondary Outcome: Time to Sustained Clinical Recovery After New Coronavirus Disease COVID-19.
Description: Sustained clinical recovery is a sustained improvement of clinical symptoms for at least 4 consecutive days. The day of improvement is considered the first of these 4 days.
  Criteria for improvement of clinical symptoms (according to the scoring system "Assessment of 14 Common COVID-19-Related Symptoms") are defined as follows:
  * a score of 1 or 0 (for stuffy or runny nose, sore throat, low energy or tiredness, muscle or body aches, headache, chills or shivering, feeling hot or feverish, nausea, diarrhea);
  * a score 0 (for shortness of breath/difficulty breathing and vomiting);
  * a score no more than 2 (for cough);
  * no new symptoms with a score of 1 or 0;
  * axillary temperature ≤37.3°С.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 381 | 389
day | 4.5 (2.4) | 5.8 (4.7)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Mean differences (Raphamin vs. Placebo) were compared; Test type: Superiority; p = 0.0025, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance is set to 0.005

3. Secondary Outcome: Percentage of Hospitalized Patients
Description: Based on the medical records.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
Participants | 0 | 0

4. Other Pre Specified Outcome: Time to COVID-19 Progression to a More Severe Form
Description: Severity of COVID-19 will be assessed in accordance with the criteria presented in the current edition of the clinical recommendations of the Ministry of Health of the Russian Federation "Prevention, diagnosis and treatment of a new coronavirus infection (COVID-19)".
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 59 | 89
day | 1.6 (0.8) | 2.4 (3.9)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Mean differences (Raphamin vs. Placebo) were compared; Test type: Superiority; p = 0.2607, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Percentage of Patients With Negative PCR Test for SARS-CoV-2
Description: Number of patients with a negative PCR test result for SARS-CoV-2 on days 6 and 10 of observation. Based on the medical records.
Time Frame: On days 6 and 10
Population: In accordance with protocol only PCR positive participants were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 102 | 95
Participants
  Day 6 | 68 | 66
  Day 10 | 93 | 89
Statistical Analysis 1: Comparison: Raphamin vs Placebo; This analysis applies to "Day 6" row; Test type: Superiority; p = 0.7601, Fisher Exact
Statistical Analysis 2: Comparison: Raphamin vs Placebo; This analysis applies to "Day 10" row; Test type: Superiority; p = 0.7685, Fisher Exact

6. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: The presence of adverse events. Based on medical records.
Time Frame: From day 1 to day 6
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
Participants | 29 | 46
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.052, Fisher Exact

7. Other Pre Specified Outcome: Severity of AEs
Description: The intensity (severity) of adverse events. Based on medical records.
Time Frame: From day 1 to day 6
Measure: Number; unit: Number of AE
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 29 | 46
Number of AE
  Mild | 25 | 43
  Moderate | 14 | 18
  Severe | 2 | 0
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.19, Fisher Exact

8. Other Pre Specified Outcome: Causal Relationship of AEs to the Sudy Drug
Description: The causal relationship to the study drug of adverse events. Based on medical records.
Time Frame: From day 1 to day 6
Measure: Number; unit: Number of AEs
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 29 | 46
Number of AEs
  No relation | 39 | 52
  Probable | 1 | 0
  Possible | 1 | 2
  Doubtful | 0 | 6
  Certain | 0 | 1
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.54, Fisher Exact

9. Other Pre Specified Outcome: Outcome of AEs
Description: The outcome of adverse events. Based on medical records.
Time Frame: From day 1 to day 6
Measure: Number; unit: Number of AEs
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 29 | 46
Number of AEs
  Recovery/resolution | 23 | 40
  Incomplete recovery/ resolution | 5 | 6
  No recovery/resolution | 1 | 0
  Unknown | 12 | 15
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.10, Fisher Exact

10. Other Pre Specified Outcome: Changes in Vital Signs: Pulse Rate/Heart Rate in Beats Per Minute (Bpm)
Description: The outcome measure is based on the medical records. The patient's heart rate (heart rate) is measured by the physician in visits 1, 3 and 4 (on days 1 and 6).
Time Frame: On Visit 1 (day 1), Visit 3 (day 6), Visit 4 (day10)
Measure: Mean (Standard Deviation); unit: Bpm
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
Bpm
  Visit 1 | 81.7 (10.4) | 81.9 (10.5)
  Visit 3 | 73.9 (6.3) | 74.4 (6.4)
  Visit 4 | 72.6 (6.0) | 73.2 (5.8)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.92, ANOVA — The p-value associated with "treatment*visit" interaction of pulse rate (heart rate) from Visit 1 to 4 between Raphamin and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

11. Other Pre Specified Outcome: Changes in Vital Signs: Respiration Rate/Breathing Rate in Breaths Per Minute
Description: Outcome Measure is based on the medical records. The patient's respiration rate (breathing rate) is measured by physician in visits 1, 3 and 4 (on days 1 and 6).
Time Frame: On Visit 1 (day 1), Visit 3 (day 6), Visit 4 (day10)
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
Breaths per minute
  Visit 1 | 17.1 (1.4) | 17.2 (1.5)
  Visit 3 | 16.6 (1.2) | 16.5 (1.4)
  Visit 4 | 16.4 (1.3) | 16.4 (1.3)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.44, ANOVA — The p-value associated with "treatment*visit" interaction of respiration rate (breathing rate) from Visit 1 to 4 between Raphamin and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

12. Other Pre Specified Outcome: Changes in Vital Signs: Capillary Blood Oxygen Saturation (SpO2)
Description: Outcome Measure is based on the medical records. The patient's capillary blood oxygen saturation (SpO2) is measured by physician in visits 1, 3 and 4 (on days 1 and 6).
Time Frame: On Visit 1 (day 1), Visit 3 (day 6), Visit 4 (day10)
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
percentage of oxygen
  Visit 1 | 97.8 (0.9) | 97.8 (0.8)
  Visit 3 | 98.3 (0.8) | 98.3 (0.8)
  Visit 4 | 98.4 (0.8) | 98.5 (0.8)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.90, ANOVA — The p-value associated with "treatment*visit" interaction of SpO2 from Visit 1 to 4 between Raphamin and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

13. Other Pre Specified Outcome: Changes in Vital Signs: Blood Pressure in Units of Millimeters of Mercury (mmHg)
Description: Outcome Measure is based on the medical records. The patient's blood pressure is measured by the physician in visits 1, 3 and 4 (on days 1 and 6).
Time Frame: On Visit 1 (day 1), Visit 3 (day 6), Visit 4 (day10)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
mmHg
  SBP/Visit 1 | 122.1 (9.5) | 122.1 (9.9)
  SBP/Visit 3 | 121.8 (8.3) | 121.2 (8.2)
  SBP/Visit 4 | 121.1 (7.6) | 121.2 (7.9)
  DBP/Visit 1 | 76.9 (6.8) | 76.8 (7.4)
  DBP/Visit 3 | 76.5 (6.2) | 76.3 (6.2)
  DBP/Visit 4 | 76.2 (6.0) | 76.1 (6.3)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.30, ANOVA — The p-value associated with "treatment*visit" interaction of SBP from Visit 1 to 4 between Raphamin and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.94, ANOVA — The p-value associated with "treatment*visit" interaction of DBP from Visit 1 to 4 between Raphamin and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

14. Other Pre Specified Outcome: Percentage of Patients With Clinically Significant Abnormal Laboratory Tests
Description: Measure is based on the Hematology, blood chemistry, and urinalysis parameters, which are beyond the reference values at the end of treatment.
Time Frame: On Visit 1 (day 1) and Visit 3 (day 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 382 | 389
Participants | 13 | 16

ADVERSE EVENTS:
Time Frame: Registration of AEs begins after the first dose of study drug and continues throughout the entire period of study therapy - 28 days.
Arm/Group | Raphamin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/382 | 0/389
Serious Adverse Events (participants affected / at risk) | 1/382 | 0/389
Other Adverse Events (participants affected / at risk) | 29/382 | 46/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raphamin (N=382) | Placebo (N=389)
Worsening of atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Worsening of persistent atrial fibrillation (symptoms of chest pain, palpitations, loss of consciousness from 22.11.2022). Hospitalized.
Complicated fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Closed, fragmented fracture of the fibula in the lower third of the left shin with displacement.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raphamin (N=382) | Placebo (N=389)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) — Without further clarification
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) — Without further clarification
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1)
Exacerbation of hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting urge (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0)
Maxillary sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis caused by herpes simplex virus (Infections and infestations) | 0 (0) | 1 (1)
Sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Exacerbation of chronic pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Recurrent urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Etmoiditis (Infections and infestations) | 0 (0) | 1 (1)
Protein in urine (Investigations) | 0 (0) | 1 (1)
Presence of ketone bodies in urine (Investigations) | 0 (0) | 1 (1)
Abnormal Physical Examination Results (Investigations) | 1 (1) | 1 (1)
Abnormal blood count (Investigations) | 0 (0) | 1 (1)
Increased blood pressure (Investigations) | 1 (1) | 2 (2) — Without further clarification
Increased ALT (Investigations) | 0 (0) | 1 (1)
Increased protein levels in urine (Investigations) | 1 (1) | 0 (0)
Increased bilirubin (Investigations) | 0 (0) | 1 (1)
Increased urinary glucose (Investigations) | 0 (0) | 1 (1)
Increased creatinine (Investigations) | 0 (0) | 1 (1)
Increased total bilirubin (Investigations) | 0 (0) | 2 (2)
Increased C-reactive protein (Investigations) | 0 (0) | 3 (3)
Increased transaminases (Investigations) | 1 (1) | 3 (3)
Increased eosinophil count (Investigations) | 1 (1) | 0 (0)
Increased neutrophil levels (Investigations) | 1 (1) | 0 (0)
Low blood pressure (Investigations) | 1 (1) | 0 (0)
Decrease in general clinical blood test values (Investigations) | 0 (0) | 1 (1)
Haematocrit reduction (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Decrease in general bilirubin levels (Investigations) | 0 (0) | 1 (1)
Decreased platelet count (Investigations) | 0 (0) | 1 (1)
Increased percentage of lymphocytes (Investigations) | 1 (1) | 0 (0)
Decreased percentage of lymphocytes (Investigations) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Without further clarification
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Generalized itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itchy face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching, cutaneous (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Itchy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Increased sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash on the face skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia unspecified (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Without further clarification
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Without further clarification
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper limb myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lumbago (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) — Without further clarification
Headache in the occipital region (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radicular pain (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Tingling sensation in the eyelids (Eye disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Exacerbation of chronic cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arterial hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
General malaise (General disorders) | 0 (0) | 1 (1)
Bruised finger (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT05364671/Prot_SAP_000.pdf